CLINICAL TRIAL: NCT02851290
Title: Effect of Caudal and Penile Block on Hypospadias Repair Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Nicolette Janzen, Assistant Professor Pediatric Urology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-38540
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Hypospadias
Keywords: Hypospadias; Caudal block; Dorsal penile nerve block; Anesthesia; Urethrocutaneous fistula; Urethral stricture; Meatal stenosis; Glanular dehiscence
MeSH Terms: conditions — Hypospadias; Urethral Stricture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caudal block (Experimental): Local anesthetic will be administered into the caudal space
  Interventions: Procedure: Caudal block anesthesia
- Dorsal penile nerve block (Active Comparator): Local anesthetic will be administered around the dorsal penile nerve
  Interventions: Procedure: Dorsal penile nerve block anesthesia

INTERVENTIONS:
Procedure: Caudal block anesthesia — After induction of general anesthesia, a caudal block will be performed using 0.75-1 mL/kg of 0.2% ropivacaine without epinephrine
  Arms: Caudal block
Procedure: Dorsal penile nerve block anesthesia — After induction of general anesthesia, a dorsal penile nerve block will be performed using 0.75-1 mL/kg of 0.2% ropivacaine without epinephrine
  Arms: Dorsal penile nerve block

SUMMARY:
Hypospadias is one of the most common genitourinary (GU) malformations, seen in approximately 1 of 250 male live births. Common methods of local anesthesia administration for hypospadias surgery include caudal and dorsal penile nerve blocks. While both methods are known to be effective with minimal risk, the effect on post-operative complications is not well-established. The purpose of this randomized controlled trial is to evaluate if caudal versus dorsal penile nerve block results in higher rates of post-operative complications.

DETAILED DESCRIPTION:
Hypospadias is a one of the most common genitourinary (GU) malformations, seen in approximately 1 of 250 male live births, characterized by proximal location of the urethral meatus, dorsal hooded foreskin with incomplete ventral fusion, and ventral curvature of the penis. Hypospadias repair includes several standard steps including urethroplasty, mobilization of adjacent flaps for urethroplasty coverage, rotation of penile skin flaps and circumcision. In order for the surgeon to operate in a clean and relatively bloodless field, tourniquets and local epinephrine injection have been used. In a rabbit hypospadias repair model, the authors used both tourniquet and local epinephrine infiltration to maintain a clear surgical field, and showed increased apoptotic urethral myocytes on TUNNEL assay and collagen deposition in the epinephrine cohort. The study also showed structural changes in the mitochondria on scanning electron microscopy in the epinephrine cohort. This is the only hypospadias study demonstrating pathologic changes in the urethra after tourniquet or epinephrine injection. While single stage hypospadias surgical techniques have standardized significantly over the two decades, surgical complications can still occur in up to 28% of patients. Complications include urethrocutaneous fistulas, meatal stenosis, glans dehiscence, urethral strictures, and urethral diverticulum. Risk factors for hypospadias surgical complications have been extensively published and include: proximal urethral location, previous operation, glans width <14 mm, no urethroplasty coverage layers, surgeon learning curve, and age <4 years old.

The majority of hypospadias surgical complications need to be revised surgically and this results in significant financial and emotional burden for the family. The financial impact of hypospadias visits, repairs, and reoperations on society is largely unknown. A single study in 2000 noted that $16.6 million was spent on operative and outpatient hypospadias care and 17,000 total outpatient hypospadias visits were made that year. No recent studies are available and the cost to the patient per surgery and per surgical complication repair is also unknown. Multiple objective hypospadias surgical questionnaires have been developed to characterize postoperative appearance of the skin, meatus, urinary stream, and presence of fistula. These studies have only been validated by the same institution and data correlating questionnaire scores to complications is sparse.

Penile sensation is derived primarily from the dorsal nerve of the penis. Ventrally there is some innervation to the frenulum that is derived from the perineal nerve branches. The dorsal nerve of the penis is a branch of the pudendal nerve which is supplied from sacral nerves. Common methods for penile block, which are performed by the hypospadias surgeon, include dorsal nerve penile block (DNPB) or penile ring block. The DNPB involves infiltration of local anesthetic using a short beveled needle in the subpubic location at the 10 and 2 o'clock positions such that the dorsal nerve of the penis is blocked as it enters the base of the penis. The penile ring block is performed by infiltration of local anesthetic in the subcutaneous tissue at the base of the penis. One prospective study showed that DNPB was significantly better than ring block. Success rates of DNPB have been noted to be anywhere from 90-100% in children undergoing circumcision. Complications from DNPB are exceptionally rare at <0.1% including hematoma and local tissue edema.

Caudal block is a commonly performed regional block by anesthesiologists for hypospadias surgery. It involves blockade of the same nerve pathway described above, at a more proximal location, by infiltration of the caudal epidural space through the sacral hiatus. The procedure is performed usually in the lateral position. Anatomic landmarks are defined by an equilateral triangle formed by the bilateral posterior superior iliac spines, and the sacral hiatus. Initially a short beveled needle or small gauge angiocatheter is inserted into the sacral hiatus at a 45 degree angle and then once a "pop" is heard, the angle is "dropped" to 0 degrees and the needle is advanced. Aspiration is performed and in the absence of cerebrospinal fluid or blood, a local anesthetic is injected. Complications are exceptionally rare at the rate of <0.003% and include local anesthetic toxicity, neurological injury or infection and success rates of up to 96% have been reported.

Penile physiology and blood flow parameters after DNPB and caudal block are largely unknown. Very few studies show the effects of distal organ perfusion after regional blockade. One study looking at children undergoing caudal block for urologic procedures found that caudal block using 1.5 ml/kg of 0.15% ropivicaine increased the dorsalis pedis arterial parameters: increased peak velocity 24%, volume flow 76%, arterial diameter 20%. The authors proposed a sympatholytic mechanism as the reason for these physiologic changes. Another randomized controlled trial primarily looking at post-operative pain outcomes in hypospadias repair patients also found increased penile volumes of 27% in the caudal block arm, with the proposed mechanism also being sympatholytic. Finally, there have been case reports in which the sympatholytic effects of caudal blocks are used to treat glans ischemia after circumcision.

Penile analgesia after caudal block is approximately equal to that of DNPB. A meta-analysis of the circumcision analgesia literature, analyzing over 700 patients showed analgesic equivalence of caudal versus parenteral analgesia. Also in the meta-analysis, caudal block was found to be equivalent to DNPB with increased motor blockade found in the caudal block arm. One randomized controlled trial assessing analgesia requirements in children undergoing hypospadias repair after caudal block and penile block found that penile block resulted in superior pain control. However, another randomized controlled trial found that caudal block resulted in superior pain control as compared to penile block. After either bock, there are usually no significant alterations in mean arterial pressure.

Recently, the association between caudal block and hypospadias surgical complications has been theorized and has drawn international interest amongst pediatric urologists and anesthesiologists. A randomized controlled trial of 54 distal hypospadias repair patients, half assigned to caudal block and half to penile block, showed that all urethrocutaneous fistulas were seen in the caudal block arm. Even though the primary outcome was post-operative pain control between the groups, the authors theorized that caudal blocks lead to sympathetic blockade, penile engorgement, tissue edema, and increased hypospadias surgical complications. A nested case control series comparing 45 fistulas and 90 controls showed no association between fistulas and caudal block. The authors found fistula to be associated with proximal urethral location, penile epinephrine injection, and longer operative times. Unpublished data presented at the 2015 American Urologic Association in New Orleans by Routh et al. showed that in a retrospective single surgeon series of 452 primary hypospadias repair patients, half which had caudal block and half which had penile block, caudal blockade was highly associated with hypospadias surgical complications even after adjusting for operative time (OR 3.9 (1.3-12.1)); p= 0.0008. This is the only study to date that has been powered appropriately to assess the association between caudal block and hypospadias complications. Thus, there is clinical equipoise regarding the utilization of caudal block versus penile block for post-operative pain control and also in minimizing surgical complications in hypospadias repair.

ELIGIBILITY:
Inclusion criteria:

* Age 4 months to 4 years
* ASA score I and II
* Primary hypospadias repair in one stage including distal, midshaft, and proximal repairs

Exclusion criteria:

* Age <4 months or >4 years
* ASA score >II
* Genetic syndromes
* Previous hypospadias operations
* Staged hypospadias repair operations
* Spinal dysraphism or other contraindications to caudal block
* Infection at the block site
* Refusal of consent by the parents
* Unwillingness of the anesthesiologist or surgeon to participate

Ages: 4 Months to 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2016-07; Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Post-operative hypospadias repair complications | 24 months post-operatively
  Post-operative follow-up to evaluate for post-operative complications including urethrocutaneous fistula, glans dehiscence, meatal stenosis, and urethral stricture

SECONDARY OUTCOMES:
Post-operative hypospadias repair pain | 1 hour post-operatively
  Post-operative pain will be assessed using the FLACC scale (faces, legs, activity, cry and consolability scale)
Caudal block-related complications | 1 hour post-operatively
  Complications related to caudal block
Dorsal penile nerve block-related complications | 1 hour post-operatively
  Complications related to dorsal penile nerve block

CONTACTS AND LOCATIONS:
Overall Officials: Nicolette K Janzen, MD, Principal Investigator — Texas Children's Hospital/Baylor College of Medicine; Kara Toman, MPH, Study Director — Texas Children's Hospital/Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No